CLINICAL TRIAL: NCT01500018
Title: A Single-center, Single-dose, Double-blind, Randomized, Placebo- and Active-controlled Crossover Study to Evaluate the Abuse Potential of TC-5214 in Healthy Recreational Polydrug Users
Brief Title: Study in Healthy Recreational Polydrug Users to Measure the Abuse Potential of TC-5214
Acronym: TC-5214
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to withdraw.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D4130C00022
Record Dates: First submitted 2011-12-06; First posted 2011-12-26 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Drug Abuse; Healthy
Keywords: Phase I; healthy recreational polydrug users; abuse liability; TC-5214; Single dose crossover study to evaluate the abuse potential of TC-5214
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ketamine; Phentermine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (14):
- Crossover Treatment Sequence 1 (Experimental): Period 1: Placebo, Period 2: Phentermine 45 mg, Period 3: Phentermine 90 mg, Period 4: Ketamine 100 mg, Period 5: TC-5214 2 mg, Period 6: TC-5214 8 mg, Period 7: TC-5214 16 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 2 (Experimental): Period 1: Phentermine 45 mg, Period 2: Ketamine 100 mg , Period 3: Placebo, Period 4: TC-5214 8 mg , Period 5: Phentermine 90 mg, Period 6: TC-5214 16 mg, Period 7: TC-5214 2 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 3 (Experimental): Period 1: Ketamine 100 mg, Period 2: TC-5214 8 mg, Period 3: Phentermine 45 mg, Period 4: TC-5214 16 mg, Period 5: Placebo, Period 6: TC-5214 2 mg, Period 7: Phentermine 90 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 4 (Experimental): Period 1: TC-5214 8 mg, Period 2: TC-5214 16 mg, Period 3: Ketamine 100 mg, Period 4: TC-5214 2 mg, Period 5: Phentermine 45 mg , Period 6: Phentermine 90 mg, Period 7: Placebo
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 5 (Experimental): Period 1: TC-5214 16 mg, Period 2: TC-5214 2 mg, Period 3: TC-5214 8 mg, Period 4: Phentermine 90 mg, Period 5: Ketamine 100 mg, Period 6: Placebo , Period 7: Phentermine 45 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 6 (Experimental): Period 1: TC-5214 2 mg, Period 2: Phentermine 90 mg, Period 3: TC-5214 16 mg, Period 4: Placebo, Period 5: TC-5214 8 mg, Period 6:Phentermine 45 mg , Period 7: Ketamine 100 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 7 (Experimental): Period 1: Phentermine 90 mg, Period 2: Placebo, Period 3: TC-5214 2 mg, Period 4: Phentermine 45 mg, Period 5: TC-5214 16 mg, Period 6: Ketamine 100 mg, Period 7: TC-5214 8 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 8 (Experimental): Period 1: TC-5214 16 mg, Period 2: TC-5214 8 mg, Period 3: TC-5214 2 mg, Period 4: Ketamine 100 mg, Period 5: Phentermine 90 mg, Period 6: Phentermine 45 mg, Period 7: Placebo
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 9 (Experimental): Period 1: TC-5214 2 mg, Period 2: TC-5214 16 mg, Period 3: Phentermine 90 mg, Period 4: TC-5214 8 mg, Period 5: Placebo, Period 6: Ketamine 100 mg, Period 7:
  Phentermine 45 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 10 (Experimental): Period 1: Phentermine 90 mg, Period 2: TC-5214 2 mg, Period 3: Placebo, Period 4: TC-5214 16 mg Ketamine 100 mg, Period 5: Phentermine 45 mg, Period 6: TC-5214 8 mg, Period 7: TC-5214 2 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 11 (Experimental): Period 1: Placebo, Period 2: Phentermine 90 mg, Period 3:Phentermine 45 mg, Period 4: TC-5214 2 mg, Period 5: Ketamine 100 mg, Period 6: TC-5214 16 mg, Period 7: TC-5214 8 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 12 (Experimental): Period 1: Phentermine 45 mg, Period 2: Placebo, Period 3: Ketamine 100 mg, Period 4:Phentermine 90 mg, Period 5: TC-5214 8 mg, Period 6: TC-5214 2 mg, Period 7: TC-5214 16 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 13 (Experimental): Period 1: Ketamine 100 mg, Period 2: Phentermine 45 mg, Period 3: TC-5214 8 mg, Period 4: Placebo, Period 5: TC-5214 16 mg, Period 6: Phentermine 90 mg, Period 7: TC-5214 2 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine
- Crossover Treatment Sequence 14 (Experimental): Period 1: TC-5214 8 mg, Period 2: Ketamine 100 mg, Period 3: TC-5214 16 mg, Period 4: Phentermine 45 mg, Period 5: TC-5214 2 mg, Period 6: Placebo, Period 7: Phentermine 90 mg
  Interventions: Drug: TC-5214; Drug: TC-5214 Placebo; Drug: Ketamine; Drug: Phentermine

INTERVENTIONS:
Drug: TC-5214 — Single oral dose of 2 mg
Drug: TC-5214 Placebo — Single oral dose
Drug: Ketamine — Single oral dose of 100 mg
Drug: Phentermine — Single oral dose of 45 mg
Drug: TC-5214 — Single oral dose of 8 mg
Drug: TC-5214 — Single oral dose of 16 mg
Drug: Phentermine — Single oral dose of 90 mg

SUMMARY:
This is a single dose, crossover study to assess the abuse potential of TC-5214 compared to placebo, ketamine, and phentermine in healthy recreational polydrug users.

DETAILED DESCRIPTION:
A Single-center, Single-dose, Double-blind, Randomized, Placebo- and Active-controlled Crossover Study to Evaluate the Abuse Potential of TC-5214 in Healthy Recreational Polydrug Users.

ELIGIBILITY:
Inclusion Criteria:

* Current recreational polydrug users with experience with at least 2 drug classes of abuse.
* At least 10 lifetime uses of stimulants drugs (eg, amphetamine, cocaine, methamphetamine) and 10 lifetime occasions of recreational use of psychedelic drugs (eg, cannabis, ketamine, dextromethorphan, PCP, MDMA [ecstasy], LSD, mesacline, or psilocybin).
* Recreational use of other classes of drugs is permitted, including opioids (eg, codeine, morphine, or heroin), minor tranquilizers, or sedatives (eg, benzodiazepines or barbiturates).
* Male or female volunteers aged 18 to 55, inclusive with a body mass index (BMI) within the range of 19.0 to 33.0 kg/m2, inclusive, and a minimum weight of 50.0 kg at screening.
* Must pass qualification phase eligibility criteria.

Exclusion Criteria:

* Self-reported history of drug or alcohol dependence (except caffeine) in the past 12 months, including subjects who have ever been in a drug rehabilitation program (other than treatment for smoking cessation).
* Unwillingness or inability to abstain from recreational drug use for the duration of the study from screening until follow-up.
* Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening.
* Any significant unstable hepatic, renal, pulmonary, cardiovascular, ophthalmologic, neurologic, or any other medical conditions that might confound the study or put the volunteer at greater risk during study participation.
* Currently smoking more than 20 cigarettes (or 2 cigars) per day, and/or unwillingness to abstain from smoking for durations of at least 12 hours.
* Use of tobacco cessation product within 1 month (eg, nicotine substitution products, bupropion, etc).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Momentary Drug Liking VAS maximum effect (Emax) | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "At this moment, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking". The maximum value recorded is chosen.

SECONDARY OUTCOMES:
Momentary Drug Liking VAS minimum effect (Emin) | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "At this moment, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking" The minimum value recorded is chosen.
Drug Liking VAS time-weighted mean (TWmean) | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "At this moment, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking". Time weighted average score is calculated.
Overall Drug Liking VAS maximum effect ( Emax) | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "Overall, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking". The maximum value recorded is chosen.
Overall Drug Liking VAS (Emin) | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "Overall, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking". The minimum value recorded is chosen
Overall Drug Liking VAS 10-hour mean score | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8 and 10 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "Overall, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking". The mean value is calculated.
Overall Drug Liking VAS 24-hour mean score | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "Overall, my liking for this drug is" with anchor points "0: Strong disliking" and "100: Strong liking". The mean value is calculated.
Take Drug Again VAS Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I would take this drug again" with anchor points "0: Definitely not" and "100: Definitely so". The maximum value recorded is chosen.
Take Drug Again VAS 10-hour mean score | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8 and 10 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I would take this drug again" with anchor points "0: Definitely not" and "100: Definitely so". The mean value is calculated
Take Drug Again VAS 24-hour mean score | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I would take this drug again" with anchor points "0: Definitely not" and "100: Definitely so". The mean value is calculated
Subjective Drug Value Emax | 10 and 24 hours post dose
  The SDV is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between the drug administered and different monetary values.
Subjective Drug Value 10 hour mean score | 10 hours post dose
  The SDV is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between the drug administered and different monetary values
Subjective Drug 24 hour mean scores | 10 and 24 hours post dose
  The SDV is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between the drug administered and different monetary values
High VAS Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I am feeling high" with anchor points "0: Definitely not" and "100: Definitely so". The maximum value recorded is chosen.
High VAS TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I am feeling high" with anchor points "0: Definitely not" and "100: Definitely so". Time weighted average score is calculated
Good Effects VAS Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I can feel good drug effects" with anchor points "0: Definitely not" and "100: Definitely so". The maximum value recorded is chosen
Good Effects VAS TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I can feel good drug effects" with anchor points "0: Definitely not" and "100: Definitely so". Time weighted average score is calculated
Addiction Research Center Inventory (ARCI) euphoria scale (MBG) Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The maximum value recorded is chosen
Addiction Research Center Inventory (ARCI) euphoria scale (MBG) TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The time-weighted mean value is calculated
Bad Effects VAS Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I can feel bad drug effects" with anchor points "0: 0: Definitely not" and "100: 0: Definitely so". The maximum value recorded is chosen
Bad Effects VAS TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I can feel bad drug effects" with anchor points "0: Definitely not" and "100: Definitely so". Time weighted average score is calculated.
ARCI dysphoria scale (LSD) Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The maximum value recorded is chosen
ARCI dysphoria scale (LSD) TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The time-weighted mean value is calculated
ARCI sedation scale (PCAG) Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The maximum value recorded is chosen
ARCI sedation scale (PCAG) TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The time-weighted mean value is calculated
Alertness/Drowsiness VAS Emin (drowsiness) | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I am feeling" with anchor points "0: Very Drowsy" and "100: Very Alert". The minimum value recorded is chosen
Alertness/Drowsiness VAS TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I am feeling" with anchor points "0: Very Drowsy" and "100: Very Alert". The time weighted mean value is calculated
Any Effects VAS Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I can feel any drug effects" with anchor points "0: 0: Definitely not" and "100: 0: Definitely so". The maximum value recorded is chosen
Any Effects VAS TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Visual analogue scale from 0 to 100 mm. The statement put is: "I can feel any drug effects" with anchor points "0: 0: Definitely not" and "100: 0: Definitely so". The time-weighted mean value is calculated
Bowdle VAS Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  13 items for which the volunteer is asked to rate his/her feelings over the past 30 minutes. Each VAS will be scored from 0 to 100, with 0 reflecting "Not at all" and 100 reflecting "Extremely". The maximum value recorded is chosen
Bowdle VAS TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  13 items for which the volunteer is asked to rate his/her feelings over the past 30 minutes. Each VAS will be scored from 0 to 100, with 0 reflecting "Not at all" and 100 reflecting "Extremely". The time-weighted mean value is calculated
ARCI A scale Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The maximum value recorded is chosen
ARCI A scale TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The time-weighted mean value is calculated
ARCI Phentermine and Benzedrine Group scale (BG) Emax | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The maximum value recorded is chosen
ARCI Phentermine and Benzedrine Group scale (BG) TWmean | 0.5, 1,1.5, 2, 2.5, 3, 4, 6, 8, 10 and 24 hours post dose
  Questionnaire to assess possible addiction. The time-weighted mean value is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, Study Director — AstraZeneca Kvzmbergagatan 12, 15185,Sodertalje, Sweden; Pierre Geoffroy, MDCM, MSC, FCFP, Principal Investigator — Syneos Health; Brendan Smyth, MD, Study Director — AstraZeneca 180 Concord Pike, Wilmington,DE 19850-5437